CLINICAL TRIAL: NCT00705679
Title: Phase 2B Safety and Effectiveness Study of Tenofovir 1% Gel, Tenofovir Disproxil Fumarate Tablet and Emtricitabine/Tenofovir Disoproxil Fumarate Tablet for the Prevention of HIV Infection in Women
Brief Title: Safety and Effectiveness of TFV 1% Gel, TDF Tablets, and FTC/TDF Tablets in Preventing HIV in Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Microbicide Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MTN-003 (VOICE); 10622 (Registry Identifier: DAIDS ES); MTN-003 (Other: Microbicide Trials Network); 5U01AI068633-05 (NIH); VOICE (Other: Microbicide Trials Network)
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Results first posted 2016-02-10 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2016-02

CONDITIONS: HIV Infections
Keywords: Microbicide; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine; Tenofovir; Vaginal Creams, Foams, and Jellies; hexadecyloxypropyl 9-(2-(phosphonomethoxy)propyl)adenine

ARMS (5):
- 1 (Experimental): TDF 300 mg tablet taken orally once daily and one FTC/TDF placebo tablet taken orally once daily for 12 to 36 months
  Interventions: Drug: Emtricitabine/tenofovir disoproxil fumarate placebo; Drug: Tenofovir disoproxil fumarate
- 2 (Experimental): TDF placebo tablet taken orally once daily and one FTC 200 mg/TDF 300 mg tablet taken orally once daily for 12 to 36 months
  Interventions: Drug: Emtricitabine/tenofovir disoproxil fumarate; Drug: Tenofovir disoproxil fumarate placebo
- 3 (Experimental): TDF placebo tablet taken orally once daily and one FTC/TDF placebo tablet taken orally once daily for 12 to 36 months
  Interventions: Drug: Emtricitabine/tenofovir disoproxil fumarate placebo; Drug: Tenofovir disoproxil fumarate placebo
- 4 (Experimental): Application of tenofovir 1% vaginal gel once daily
  Interventions: Drug: Tenofovir 1% vaginal gel
- 5 (Experimental): Application of tenofovir placebo gel once daily
  Interventions: Drug: Tenofovir placebo

INTERVENTIONS:
Drug: Emtricitabine/tenofovir disoproxil fumarate — 200 mg/300 mg tablet
  Other Names: FTC/TDF; Truvada
  Arms: 2
Drug: Emtricitabine/tenofovir disoproxil fumarate placebo — placebo tablet
  Other Names: FTC/TDF placebo; Truvada placebo
  Arms: 1; 3
Drug: Tenofovir disoproxil fumarate — 300 mg tablet
  Other Names: TDF
  Arms: 1
Drug: Tenofovir disoproxil fumarate placebo — placebo tablet
  Other Names: TDF placebo
  Arms: 2; 3
Drug: Tenofovir 1% vaginal gel — 1 gm/100 ml of 1% gel
  Other Names: TFV; 9-[2-(Phosphonomethoxy)propyl]adenine
  Arms: 4
Drug: Tenofovir placebo — placebo gel
  Other Names: TFV placebo
  Arms: 5

SUMMARY:
A new approach to HIV prevention currently being studied includes the use of microbicides, substances that kill microbes. Tenofovir disoproxil fumarate (TDF) and emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) are oral, FDA-approved, anti-HIV drugs, and tenofovir gel is an experimental microbicide. The purpose of this study is to determine the safety and effectiveness of daily tenofovir 1% gel compared to a vaginal placebo gel, and the safety and effectiveness of oral TDF and oral FTC/TDF compared to an oral placebo in preventing HIV infection among women at risk for sexually transmitted infections.

DETAILED DESCRIPTION:
It is necessary to monitor both the adherence and blood levels of microbicides in order to gauge its efficacy in a study population. Utilizing an experimental microbicide (tenofovir gel) and anti-HIV drugs (TDF, FTC/TDF), this study will measure the effectiveness and safety to and blood levels of the three interventions in three regimens given to HIV uninfected women.

The expected duration of participation for each participant ranges from a minimum of 12 months to a maximum of 38 months. Study participants will be randomly assigned into one of five study groups, each with a different regimen. Group 1 participants will take one TDF tablet daily and one FTC/TDF placebo tablet daily. Group 2 participants will take one TDF placebo tablet daily and one FTC/TDF tablet daily. Group 3 participants will take one TDF placebo tablet daily and one FTC/TDF placebo tablet daily. Group 4 participants will apply tenofovir 1% gel vaginally once daily. Group 5 participants will apply tenofovir 1% placebo gel vaginally once daily.

Study visits will occur every 28 days after enrollment. Medical history, a physical exam, behavioral and adherence assessment, urine and blood collection, and counseling will occur at all visits. Blood will also be collected and archived for future research at select visits. Pharmacokinetic studies will occur at some visits. A pap smear will occur at select visits. Some participants may have hair samples collected on an optional basis at study visits every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide adequate locator information
* Sexually active, defined as having vaginal intercourse at least once in the 3 months prior to screening
* Agree to not participate in other research studies involving drugs, medical devices, or vaginal products for duration of study.
* Agree to use effective method of contraception. More information on this criterion can be found in the protocol.

Exclusion Criteria:

* HIV infected
* Known adverse reaction to any of the study products
* Known adverse reaction to latex
* Pathologic bone fracture not related to trauma
* Non-therapeutic injection drug use in the 12 months prior to screening
* Post-exposure prophylaxis for HIV exposure within 6 months prior to enrollment
* Last pregnancy outcome 42 days or less prior to enrollment
* Gynecologic or genital procedure 42 days or less prior to enrollment
* Participation in any other research study involving drugs, medical devices, or vaginal products 30 days or less prior to enrollment
* Currently using spermicide, interferon or interleukin therapy, or certain medications. More information on this criterion can be found in the protocol.
* Any significant uncontrolled active or chronic disease. More information on this criterion can be found in the protocol.
* Certain abnormal laboratory values. More information on this criterion can be found in the protocol.
* Intends to become pregnant in the 24 months after enrollment
* Plans to relocate or travel away from the study site for more than 8 consecutive weeks in the 24 months after enrollment
* Urinary tract infection
* Pelvic inflammatory disease, an STI, or reproductive tract infection requiring treatment
* Grade 2 or higher pelvic exam finding
* Any condition that, in the opinion of the investigator, would interfere with the study
* Pregnant or breastfeeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5029 (Actual)
Dates: Start 2009-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zvavahera M. Chirenje, MD, FRCOG, Study Chair — UZ-UCSF Collaborative Research Programme; Jeanne Marrazzo, MD, MPH, Study Chair — University of Washington, Division of Allergy and Infectious Disease
Locations (15):
- South Africa (11):
  - Wits Reproductive Health and HIV Institute CRS (WRHI CRS), Johannesburg, Gauteng
  - Soweto MTN CRS, Johannesburg, Gauteng
  - Overport CRS, Asherville, KwaZulu-Natal
  - Chatsworth CRS, Chatsworth, KwaZulu-Natal
  - eThekwini CRS, Durban, KwaZulu-Natal
  - Umkomaas CRS, eMkhomazi, KwaZulu-Natal
  - Tongaat CRS, Tongaat, KwaZulu-Natal
  - Verulam CRS, Verulam, KwaZulu-Natal
  - Botha's Hill CRS, Westville, KwaZulu-Natal
  - Isipingo CRS, Westville, KwaZulu-Natal
  - CAPRISA Aurum CRS, Klerksdorp
- MU-JHU Research Collaboration CRS, Kampala, Uganda
- Zimbabwe (3):
  - Seke South CRS, Chitungwiza
  - Zengeza CRS, Chitungwiza
  - Spilhaus CRS, Harare

REFERENCES:
- [Background] Mayer KH, Maslankowski LA, Gai F, El-Sadr WM, Justman J, Kwiecien A, Masse B, Eshleman SH, Hendrix C, Morrow K, Rooney JF, Soto-Torres L; HPTN 050 Protocol Team. Safety and tolerability of tenofovir vaginal gel in abstinent and sexually active HIV-infected and uninfected women. AIDS. 2006 Feb 28;20(4):543-51. doi: 10.1097/01.aids.0000210608.70762.c3. PMID 16470118
- [Background] Rosen RK, Morrow KM, Carballo-Dieguez A, Mantell JE, Hoffman S, Gai F, Maslankowski L, El-Sadr WM, Mayer KH. Acceptability of tenofovir gel as a vaginal microbicide among women in a phase I trial: a mixed-methods study. J Womens Health (Larchmt). 2008 Apr;17(3):383-92. doi: 10.1089/jwh.2006.0325. PMID 18328009
- [Derived] Chirenje ZM, Gundacker HM, Richardson B, Rabe L, Gaffoor Z, Nair GL, Mirembe BG, Piper JM, Hillier S, Marrazzo J. Risk Factors for Incidence of Sexually Transmitted Infections Among Women in a Human Immunodeficiency Virus Chemoprevention Trial: VOICE (MTN-003). Sex Transm Dis. 2017 Mar;44(3):135-140. doi: 10.1097/OLQ.0000000000000568. PMID 28178109
- [Derived] Moodley J, Naidoo S, Moodley J, Ramjee G. Sharing of Investigational Drug Among Participants in the Voice Trial. AIDS Behav. 2016 Nov;20(11):2709-2714. doi: 10.1007/s10461-016-1414-x. PMID 27146827
- [Derived] van der Straten A, Brown ER, Marrazzo JM, Chirenje MZ, Liu K, Gomez K, Marzinke MA, Piper JM, Hendrix CW; MTN-003 VOICE Protocol Team for Microbicide Trials Network. Divergent adherence estimates with pharmacokinetic and behavioural measures in the MTN-003 (VOICE) study. J Int AIDS Soc. 2016 Feb 4;19(1):20642. doi: 10.7448/IAS.19.1.20642. eCollection 2016. PMID 26850270
- [Derived] Noguchi LM, Richardson BA, Baeten JM, Hillier SL, Balkus JE, Chirenje ZM, Bunge K, Ramjee G, Nair G, Palanee-Phillips T, Selepe P, van der Straten A, Parikh UM, Gomez K, Piper JM, Watts DH, Marrazzo JM; VOICE Study Team. Risk of HIV-1 acquisition among women who use diff erent types of injectable progestin contraception in South Africa: a prospective cohort study. Lancet HIV. 2015 Jul;2(7):e279-87. doi: 10.1016/S2352-3018(15)00058-2. PMID 26155597
- [Derived] Dai JY, Hendrix CW, Richardson BA, Kelly C, Marzinke M, Chirenje ZM, Marrazzo JM, Brown ER. Pharmacological Measures of Treatment Adherence and Risk of HIV Infection in the VOICE Study. J Infect Dis. 2016 Feb 1;213(3):335-42. doi: 10.1093/infdis/jiv333. Epub 2015 Jun 29. PMID 26123563
- [Derived] Marrazzo JM, Ramjee G, Richardson BA, Gomez K, Mgodi N, Nair G, Palanee T, Nakabiito C, van der Straten A, Noguchi L, Hendrix CW, Dai JY, Ganesh S, Mkhize B, Taljaard M, Parikh UM, Piper J, Masse B, Grossman C, Rooney J, Schwartz JL, Watts H, Marzinke MA, Hillier SL, McGowan IM, Chirenje ZM; VOICE Study Team. Tenofovir-based preexposure prophylaxis for HIV infection among African women. N Engl J Med. 2015 Feb 5;372(6):509-18. doi: 10.1056/NEJMoa1402269. PMID 25651245

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women were recruited from September 2009 through June 2011 from 15 sites in South Africa, Uganda, and Zimbabwe.
Pre-assignment Details: 12,320 women were assessed for eligibility and 7,291 were excluded for various reasons, including 2,308 women who were HIV-positive. 5,029 women were randomized.
Groups:
- Oral TDF: TDF 300 mg tablet taken orally once daily and one FTC/TDF placebo tablet taken orally once daily for 12 to 36 months
  Emtricitabine/tenofovir disoproxil fumarate placebo: placebo tablet
  Tenofovir disoproxil fumarate: 300 mg tablet
- Oral TDF-FTC: TDF placebo tablet taken orally once daily and one FTC 200 mg/TDF 300 mg tablet taken orally once daily for 12 to 36 months
  Emtricitabine/tenofovir disoproxil fumarate: 200 mg/300 mg tablet
  Tenofovir disoproxil fumarate placebo: placebo tablet
- Oral Placebo: TDF placebo tablet taken orally once daily and one FTC/TDF placebo tablet taken orally once daily for 12 to 36 months
  Emtricitabine/tenofovir disoproxil fumarate placebo: placebo tablet
  Tenofovir disoproxil fumarate placebo: placebo tablet
- TFV Gel: Application of tenofovir 1% vaginal gel once daily
  Tenofovir 1% vaginal gel: 1 gm/100 ml of 1% gel
- Gel Placebo: Application of tenofovir placebo gel once daily
  Tenofovir placebo: placebo gel
Period: Overall Study
Arm/Group | Oral TDF | Oral TDF-FTC | Oral Placebo | TFV Gel | Gel Placebo
Started | 1007 | 1003 | 1009 | 1007 | 1003
Completed | 942 | 864 | 894 | 927 | 934
Not Completed | 65 | 139 | 115 | 80 | 69
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 3 | 2 | 1
Not completed — Lost to Follow-up | 32 | 60 | 44 | 30 | 35
Not completed — Physician Decision | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 32 | 77 | 68 | 47 | 33

BASELINE CHARACTERISTICS:
Population: Includes all participants enrolled and randomized to a study arm
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral TDF | Oral TDF-FTC | Oral Placebo | TFV Gel | Gel Placebo | Total
Number analyzed (Participants) | 1007 | 1003 | 1009 | 1007 | 1003 | 5029
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.5 (5.1) | 25.2 (5.2) | 25.3 (5.2) | 25.3 (5.2) | 25.3 (5.1) | 25.3 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1007 | 1003 | 1009 | 1007 | 1003 | 5029
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — Response to the question: What is your ethnic group or tribe?
  participants
    Chichewa | 4 | 10 | 7 | 7 | 2 | 30
    Lombwe | 0 | 0 | 0 | 0 | 1 | 1
    Yao | 1 | 0 | 0 | 0 | 1 | 2
    Tumbuka | 0 | 1 | 1 | 0 | 1 | 3
    Other African tribe | 76 | 75 | 83 | 92 | 84 | 410
    White | 0 | 0 | 0 | 0 | 0 | 0
    Zulu | 601 | 587 | 595 | 585 | 571 | 2939
    Xhosa | 85 | 75 | 74 | 72 | 92 | 398
    Indian | 21 | 28 | 22 | 22 | 22 | 115
    Colored | 0 | 3 | 3 | 4 | 1 | 11
    Black | 64 | 64 | 65 | 65 | 64 | 322
    Bemba | 0 | 0 | 0 | 0 | 0 | 0
    Chewa | 1 | 1 | 0 | 0 | 0 | 2
    Tonga | 0 | 0 | 0 | 0 | 0 | 0
    Lozi | 0 | 0 | 0 | 0 | 0 | 0
    Shona | 123 | 108 | 111 | 111 | 117 | 570
    Ndebele | 14 | 27 | 18 | 25 | 22 | 106
    Other | 17 | 24 | 30 | 24 | 25 | 120
Region of Enrollment [Number; unit: participants] — Country at time of enrollment
  participants
    South Africa | 816 | 812 | 815 | 818 | 816 | 4077
    Uganda | 64 | 64 | 65 | 65 | 64 | 322
    Zimbabwe | 127 | 127 | 129 | 124 | 123 | 630
Some secondary school education or higher [Number; unit: participants] — Response to question: What is your highest level of education?
  participants
    Some secondary school education or higher | 924 | 929 | 926 | 920 | 923 | 4622
    Complete primary school education or lower | 82 | 74 | 83 | 85 | 79 | 403
    Missing | 1 | 0 | 0 | 2 | 1 | 4
Earns own income [Number; unit: participants] — Response to question: Do you earn an income of your own?
  participants
    Yes | 569 | 569 | 586 | 587 | 570 | 2881
    No | 438 | 434 | 423 | 420 | 432 | 2147
    Missing | 0 | 0 | 0 | 0 | 1 | 1
Live births [Mean (Standard Deviation); unit: children] — Response to question: How many children have you given birth to who were alive at birth?
  children | 1.6 (1.1) | 1.5 (1.1) | 1.5 (1.2) | 1.5 (1.1) | 1.5 (1.2) | 1.5 (1.1)
Currently married [Number; unit: participants] — Response to question: Are you currently married?
  participants
    Yes | 207 | 209 | 211 | 210 | 215 | 1052
    No | 800 | 794 | 798 | 797 | 788 | 3977
At least 2 male sex partners in the past 3 months [Number; unit: participants] — Includes primary partner and at least 1 other male partner with which the participant has had vaginal sex in the past 3 months
  participants
    Yes | 236 | 208 | 244 | 217 | 199 | 1104
    No | 761 | 782 | 754 | 779 | 793 | 3869
    No response | 10 | 13 | 11 | 11 | 11 | 56
Episodes of vaginal intercourse in the past 7 days [Mean (Standard Deviation); unit: episodes] | 2.5 (2.8) | 2.5 (3.4) | 2.5 (2.6) | 2.6 (3.6) | 2.6 (2.9) | 2.5 (3.1)
Condom use during last vaginal intercourse [Number; unit: participants]
  Yes | 763 | 760 | 742 | 768 | 733 | 3766
  No | 242 | 239 | 263 | 239 | 268 | 1251
  Missing | 2 | 4 | 4 | 0 | 2 | 12
Anal sex in the previous 3 months [Number; unit: participants] — A response of 1 or more to the question: In the past 3 months how many times have you had anal sex?
  participants
    Yes | 164 | 175 | 174 | 179 | 176 | 868
    No | 827 | 812 | 823 | 814 | 810 | 4086
    Missing | 16 | 16 | 12 | 14 | 17 | 75
Injectable contraception use [Number; unit: participants] — Response to question: What method(s) of contraception/family planning is the participant currently using? (Participant could indicate more than one method.)
  participants
    Yes | 709 | 723 | 700 | 707 | 726 | 3565
    No | 298 | 280 | 309 | 300 | 277 | 1464
Oral pills contraception [Number; unit: participants] — Response to question: What method(s) of contraception/family planning is the participant currently using? (Participant could indicate more than one method.)
  participants
    Yes | 226 | 223 | 238 | 238 | 215 | 1140
    No | 781 | 780 | 771 | 769 | 788 | 3889
Infection by Chlamydia trachomatis [Number; unit: participants] — Testing was performed with the use of a strand-displacement amplification assay
  participants
    Yes | 122 | 117 | 127 | 116 | 129 | 611
    No | 884 | 886 | 882 | 891 | 874 | 4417
    Missing | 1 | 0 | 0 | 0 | 0 | 1
Infection by Neisseria gonorrhoeae [Number; unit: participants] — Testing was performed with the use of a strand-displacement amplification assay
  participants
    Yes | 42 | 27 | 34 | 24 | 36 | 163
    No | 964 | 976 | 975 | 983 | 967 | 4865
    Missing | 1 | 0 | 0 | 0 | 0 | 1
Infection by Trichomonas vaginalis [Number; unit: participants] — Testing was performed with the use of the OSOM Trichomonas Rapid Test
  participants
    Yes | 68 | 54 | 66 | 62 | 51 | 301
    No | 939 | 948 | 943 | 943 | 949 | 4722
    Missing | 0 | 1 | 0 | 2 | 3 | 6
Syphilis infection [Number; unit: participants] — Testing was performed with the use of a rapid plasma reagin screening test followed by a confirmatory microhemagglutinin assay
  participants
    Yes | 12 | 15 | 16 | 14 | 11 | 68
    No | 994 | 988 | 993 | 993 | 992 | 4960
    Missing | 1 | 0 | 0 | 0 | 0 | 1
HSV-2 infection [Number; unit: participants] — HSV-2 seropositivity was determined with the use of the HerpeSelect 2 enzyme immunoassay at the time of enrollment; an index value of 3.5 or greater was considered to be a positive result.
  participants
    Yes | 482 | 449 | 455 | 438 | 465 | 2289
    No | 520 | 548 | 551 | 566 | 531 | 2716
    Missing | 5 | 6 | 3 | 3 | 7 | 24
Bacterial vaginosis infection [Number; unit: participants] — Bacterial vaginosis was determined by the Nugent score on Gram's staining of vaginal fluid (Nugent score 7-10).
  participants
    Yes | 422 | 410 | 401 | 397 | 393 | 2023
    No | 578 | 592 | 607 | 606 | 604 | 2987
    Missing | 7 | 1 | 1 | 4 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Person-years of Follow-up of Tenofovir 1% Gel and Vaginal Placebo Gel Arms
Description: Participants were followed for up to 30 months. Person-years measures the amount of time for each participant, in years, from the date of enrollment to the date of the first HIV-positive test result if HIV-infected during follow-up or to the date of the last HIV-negative test result on follow-up if not HIV-infected during follow-up.
Time Frame: For up to 30 months of follow-up
Population: All participants randomized except for those with no follow-up HIV testing or those determined to be HIV-positive at the time of randomization by PCR testing of plasma samples stored at the enrollment visit.
Measure: Number; unit: person-years
Groups:
- Placebo Gel: Application of placebo gel once daily Tenofovir placebo gel: placebo gel
Arm/Group | TFV Gel | Placebo Gel
Number analyzed (Participants) | 996 | 996
person-years | 1024 | 1030

2. Primary Outcome: Number of HIV-1 Infections of Tenofovir 1% Gel and Vaginal Placebo Gel Arms
Description: Participants were followed for up to 30 months. Participants were tested monthly for HIV-1 and positive rapid test results were confirmed by means of an enzyme-linked immunosorbent assay (EIA) and subsequent Western blotting (WB).
Time Frame: For up to 30 months of follow-up
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | TFV Gel | Placebo Gel
Number analyzed (Participants) | 996 | 996
participants | 61 | 70

3. Secondary Outcome: Frequency of HIV-1 Drug Resistance in Women Who Acquire HIV-1 Infection While Using Study Product
Description: The primary resistance mutations for the study were pre-defined as K65R and K70E (which confer resistance to TDF), and M184I and M184V (which confer resistance to FTC), for their potential to cause a decrease in susceptibility to the study drug. K65R, K70E, and M184I were not detected in HIV-1 from any HIV-1 seroconverters while on study product. The number of HIV-1 seroconverters while on study with the M184V resistance mutation are reported for this outcome measure.
Time Frame: Throughout study, up to 2.5 years
Population: Resistance testing was successfully completed on plasma from 301/312 HIV-1 seroconverters while on study product. 11 participants did not have a resistance result due to no stored plasma, insufficient copies of HIV-1 RNA for extraction, or PCR amplification failure.
Measure: Number; unit: participants
Arm/Group | Oral TDF | Oral TDF-FTC | Oral Placebo | TFV Gel | Gel Placebo
Number analyzed (Participants) | 58 | 55 | 60 | 60 | 69
participants
  M184V mutation | 0 | 1 | 0 | 0 | 0
  No M184V mutation | 58 | 54 | 60 | 60 | 68

4. Primary Outcome: Incidence Rate of HIV-1 Infections of Tenofovir 1% Gel and Vaginal Placebo Gel Arms
Description: This is the number of HIV-1 infections divided by the amount of person-years of follow-up time to HIV-1 infection status, multiplied by 100 (per 100 person-years).
Time Frame: For up to 30 months of follow-up
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: cases per 100 person-years
Arm/Group | TFV Gel | Placebo Gel
Number analyzed (Participants) | 996 | 996
cases per 100 person-years | 6.0 [4.6 to 7.6] | 6.8 [5.3 to 8.6]
Statistical Analysis 1: Comparison: TFV Gel vs Placebo Gel; The null hypothesis is that the active product will be no more than 25% effective. The trial was designed so that 94 events per pairwise comparison are needed to detect 55% effectiveness while ruling out a lower effectiveness of 25% with 90% power and a false-positive error rate of 0.0025; Test type: Superiority or Other; p = 0.37, Regression, Cox — The two-sided test a priori threshold for statistical significance is 0.05 against an alternative of 0% effectiveness for estimated effectiveness levels between 33.3% and 50.0%; The Cox proportional-hazards model was stratified by site; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.61 to 1.21] — A ratio less than 1 indicates a lower rate of HIV infection in the active arm compared to the placebo arm. A ratio more than 1 indicates a higher rate of HIV infection in the active arm compared to the placebo arm

5. Primary Outcome: Person-years of Follow-up of Oral TDF and Oral Placebo Arms
Description: Participants were followed for up to 30 months. Person-years measures the amount of time for each participant, in years, from the date of enrollment to the date of the first HIV-positive test result if HIV-infected during follow-up or to the date of the last HIV-negative test result on follow-up if not HIV-infected during follow-up. Note that the data for both of these arms were censored on the date when sites were asked to discontinue treatment in the oral TDF group.
Time Frame: For up to 30 months of follow-up
Population: as for outcome 1
Measure: Number; unit: person-years
Arm/Group | Oral TDF | Oral Placebo
Number analyzed (Participants) | 993 | 999
person-years | 823 | 838

6. Primary Outcome: Number of HIV-1 Infections of Oral TDF and Oral Placebo Arms
Description: as for outcome 2
Time Frame: For up to 30 months of follow-up
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Oral TDF | Oral Placebo
Number analyzed (Participants) | 993 | 999
participants | 52 | 35

7. Primary Outcome: Incidence Rate of HIV-1 Infections of Oral TDF and Oral Placebo Arms
Description: as for outcome 4
Time Frame: For up to 30 months of follow-up
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: cases per 100 person-years
Arm/Group | Oral TDF | Oral Placebo
Number analyzed (Participants) | 993 | 999
cases per 100 person-years | 6.3 [4.7 to 8.3] | 4.2 [2.9 to 5.8]
Statistical Analysis 1: Comparison: Oral TDF vs Oral Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.07, Regression, Cox — [p-value comment as in outcome 4, analysis 1]; The Cox proportional-hazards model was stratified by site; Hazard Ratio (HR) = 1.49, 95% CI 2-sided [0.97 to 2.29] — [estimate comment as in outcome 4, analysis 1]

8. Primary Outcome: Person-years of Follow-up of Oral TDF-FTC and Oral Placebo Arms
Description: as for outcome 1
Time Frame: For up to 30 months of follow-up
Population: as for outcome 1
Measure: Number; unit: person-years
Arm/Group | Oral TDF-FTC | Oral Placebo
Number analyzed (Participants) | 985 | 999
person-years | 1284 | 1308

9. Primary Outcome: Number of HIV-1 Infections of Oral TDF-FTC and Oral Placebo Arms
Description: as for outcome 2
Time Frame: For up to 30 months of follow-up
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Oral TDF-FTC | Oral Placebo
Number analyzed (Participants) | 985 | 999
participants | 61 | 60

10. Primary Outcome: Incidence Rate of HIV-1 Infections of Oral TDF-FTC and Oral Placebo Arms
Description: as for outcome 4
Time Frame: For up to 30 months of follow-up
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: cases per 100 person-years
Arm/Group | Oral TDF-FTC | Oral Placebo
Number analyzed (Participants) | 985 | 999
cases per 100 person-years | 4.7 [3.6 to 6.1] | 4.6 [3.5 to 5.9]
Statistical Analysis 1: Comparison: Oral TDF-FTC vs Oral Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.81, Regression, Cox — [p-value comment as in outcome 4, analysis 1]; The Cox proportional-hazards model was stratified by site; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.73 to 1.49] — [estimate comment as in outcome 4, analysis 1]

11. Primary Outcome: Extended Safety of Daily Tenofovir 1% Gel, Oral TDF, and Oral FTC/TDF in Women at Risk for Sexually Transmitted HIV Infection Based on Occurrence of Grade 2, 3, and 4 Adverse Events
Description: This measure describes the number of participants with elevated serum creatinine levels, the only safety outcome of concern where a significant difference was detected between an active arm and the corresponding placebo arm.
Time Frame: Throughout study, up to 2.5 years
Population: All participants randomized (intention-to-treat).
Measure: Number; unit: participants
Arm/Group | Oral TDF | Oral TDF-FTC | Oral Placebo | TFV Gel | Gel Placebo
Number analyzed (Participants) | 1007 | 1003 | 1009 | 1007 | 1003
participants | 4 | 13 | 2 | 9 | 3
Statistical Analysis 1: Comparison: Oral TDF-FTC vs Oral Placebo; Test type: Superiority or Other; p = 0.004, Fisher Exact; Two-sided Fisher's Exact Test

ADVERSE EVENTS:
Time Frame: each participant followed on study up to 2 years, 6 months
Description: Participants systematically reported any adverse experiences at monthly follow-up visits.
Arm/Group | Oral TDF | Oral TDF-FTC | Oral Placebo | TFV Gel | Gel Placebo
Serious Adverse Events (participants affected / at risk) | 17/1007 | 42/1003 | 57/1009 | 39/1007 | 26/1003
Other Adverse Events (participants affected / at risk) | 646/1007 | 740/1003 | 747/1009 | 705/1007 | 715/1003
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral TDF (N=1007) | Oral TDF-FTC (N=1003) | Oral Placebo (N=1009) | TFV Gel (N=1007) | Gel Placebo (N=1003)
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Congenital anomaly in offspring (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 3 | 1
Keratoconus (Eye disorders) | 0 | 1 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 1 | 0
Suprapubic pain (General disorders) | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 2 | 1 | 1
Bartholin's abscess (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Disseminated tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 3 | 0 | 1
Gingival abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Malaria (Infections and infestations) | 0 | 1 | 1 | 2 | 0
Meningitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Meningitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Pericarditis tuberculous (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 1 | 2 | 1 | 3
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Vulval abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Wound sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0
Electric shock (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 0
Internal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Stab wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Gliomatosis cerebri (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 1 | 4 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Meningism (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Optic neuritis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1 | 1 | 0
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 4 | 4 | 3 | 2
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0
Intrapartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Post abortion haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 4 | 2 | 1 | 2
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 5 | 1 | 1
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 0 | 0
Retained products of conception (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Depression suicidal (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 2 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Bartholin's cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Breast discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Breast enlargement (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oral TDF (N=1007) | Oral TDF-FTC (N=1003) | Oral Placebo (N=1009) | TFV Gel (N=1007) | Gel Placebo (N=1003)
Genitourinary chlamydia infection (Infections and infestations) | 105 | 144 | 154 | 100 | 107
Genitourinary tract gonococcal infection (Infections and infestations) | 26 | 46 | 45 | 40 | 32
Urinary tract infection (Infections and infestations) | 26 | 40 | 43 | 28 | 36
Vaginitis bacterial (Infections and infestations) | 31 | 41 | 41 | 32 | 43
Vulvovaginal candidiasis (Infections and infestations) | 43 | 58 | 54 | 59 | 51
Vulvovaginitis trichomonal (Infections and infestations) | 62 | 65 | 66 | 46 | 55
Alanine aminotransferase increased (Investigations) | 90 | 99 | 116 | 90 | 84
Aspartate aminotransferase increased (Investigations) | 69 | 87 | 88 | 73 | 58
Blood phosphorus decreased (Investigations) | 29 | 26 | 34 | 40 | 29
Haemoglobin decreased (Investigations) | 20 | 38 | 44 | 27 | 29
Hypophosphataemia (Metabolism and nutrition disorders) | 171 | 180 | 184 | 188 | 169
Headache (Nervous system disorders) | 32 | 39 | 44 | 23 | 30
Dysuria (Renal and urinary disorders) | 143 | 159 | 176 | 170 | 188
Pollakiuria (Renal and urinary disorders) | 16 | 39 | 41 | 30 | 34
Proteinuria (Renal and urinary disorders) | 154 | 203 | 180 | 165 | 183
Cervical dysplasia (Reproductive system and breast disorders) | 34 | 100 | 90 | 48 | 49
Menorrhagia (Reproductive system and breast disorders) | 16 | 21 | 29 | 33 | 26
Metrorrhagia (Reproductive system and breast disorders) | 29 | 55 | 50 | 48 | 51
Pelvic pain (Reproductive system and breast disorders) | 31 | 46 | 52 | 56 | 52
Vaginal discharge (Reproductive system and breast disorders) | 100 | 129 | 124 | 119 | 122
Vulvovaginal pruritus (Reproductive system and breast disorders) | 56 | 75 | 80 | 150 | 126

LIMITATIONS AND CAVEATS:
In September 2011, the oral TDF arm was discontinued for futility; in November 2011, the TFV gel and gel placebo arms were discontinued for futility. The TDF-FTC and oral placebo arms continued follow-up until the end of study in August 2012.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No